CLINICAL TRIAL: NCT00429520
Title: Prospective, Multicentre, Not Controlled Clinical Study to Investigate Efficacy and Tolerability of the Hyaluronic Acid Filler IMD1 Basic After Single Bilateral Injection for Correction of Nasolabial Folds (NLF)
Brief Title: Hyaluronic Acid Filler IMD1 Basic for Correction of Nasolabial Folds
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRZ 90026-0423/1
Record Dates: First submitted 2007-01-30; First posted 2007-01-31 (Estimated); Last update posted 2008-02-07 (Estimated); Status verified 2008-02

CONDITIONS: Nasolabial Folds

INTERVENTIONS:
Drug: Hyaluronic acid filler/IMD1 basic

SUMMARY:
Volunteers receive one injection IMD1 basic of correction of nasolabial folds and are followed-up for up to 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* main inclusion criteria: severity rating scale grade 3 or 4

Exclusion Criteria:

* main exclusion criterion: other nasolabial fold corrections within 6 months prior to study entry

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114
Dates: Start 2005-12; Study Completion 2006-12

PRIMARY OUTCOMES:
Severity rating scale assessed by independent rater

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Reinmüller, MD, Principal Investigator — Klinik am Sonnenberg, Wiesbaden, Germany
Locations (1):
- Merz Pharmaceuticals, Frankfurt, Germany